CLINICAL TRIAL: NCT00112320
Title: Randomized Trial of Pulmonary Valve Replacement in Tetralogy of Fallot
Brief Title: Comparison of Two Pulmonary Valve Replacement Methods to Treat Tetralogy of Fallot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Judith Geva, Study coordinator, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 188; P50HL074734 (NIH); P50HL074734-01 (NIH)
Record Dates: First submitted 2005-06-01; First posted 2005-06-02 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Tetralogy of Fallot; Pulmonary Valve Insufficiency; Ventricular Dysfunction, Right
Keywords: Pulmonary Valve Regurgitation; Right Ventricular Dysfunction; Heart Diseases
MeSH Terms: conditions — Tetralogy of Fallot; Pulmonary Valve Insufficiency; Ventricular Dysfunction, Right; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Standard PVR
  Interventions: Procedure: Standard PVR
- 2 (Experimental): PVR plus RV remodeling
  Interventions: Procedure: PVR plus RV remodeling

INTERVENTIONS:
Procedure: PVR plus RV remodeling — PVR and surgical RV remodeling, which includes bioprosthetic pulmonary valve insertion and resection of akinetic scarred areas on the anterior RV wall to reduce RV volume
  Arms: 2
Procedure: Standard PVR — PVR alone, which includes bioprosthetic pulmonary valve insertion and, when present, resection of right ventricular outflow tract (RVOT) aneurysm
  Arms: 1

SUMMARY:
Repair of tetralogy of Fallot (TOF), the most common form of cyanotic congenital heart disease, usually involves surgery on the outflow of the right ventricle (RV) and the pulmonary valve in order to relieve obstruction to blood flow from the RV to the lungs. This procedure often leads to regurgitation (leakage) of the pulmonary valve, which puts the burden of handling a larger than normal amount of blood flow on the RV. Over the years, that extra burden leads to enlargement of the RV and to a decrease in its function. Treatment often includes surgical insertion or replacement of a new pulmonary valve. Replacement of the damaged pulmonary valve aims to minimize the leakage and help the RV function better. This study is designed to compare two methods of how the operation (called pulmonary valve replacement [PVR]) is performed. In the first method, a new valve is inserted and only the area of the old valve is operated on; this is the standard PVR. The second method involves inserting the new valve in the same way as the standard method but, in addition, areas of the right ventricular wall that are scarred and not functioning well are removed (PVR plus right ventricular remodeling). This study will evaluate which method is more effective based on the size and function of the RV measured by cardiac magnetic resonance imaging (CMR) six months following surgery, as compared to its size and function before the operation.

DETAILED DESCRIPTION:
Background:

Surgical repair of TOF often results in chronic pulmonary regurgitation (PR) with associated RV dilatation and dysfunction. Mounting evidence indicates that PR leads to significant long-term morbidity and mortality, including arrhythmias, sudden death, and right heart failure. Using CMR, there is a high prevalence of regional dysfunction and aneurysms in the RV in patients with repaired TOF. Current standard clinical practice in patients with repaired TOF, severe PR, ventricular dysfunction, and/or clinical deterioration is to insert a bioprosthetic pulmonary valve to reduce the volume load on the RV. Although PVR can be achieved with low mortality, research has shown a persistent or worsening RV dysfunction postoperatively, despite a competent pulmonary valve. In patients with left ventricular (LV) aneurysms, surgical remodeling with aneurysm resection has been shown to improve LV mechanics. In view of the potentially deleterious effects of aneurysmal and akinetic wall segments on RV mechanics, researcher have recently modified their PVR surgical technique in selected patients to include surgical remodeling of the RV with resection of the akinetic wall segments. However, no studies have systematically compared the efficacy of PVR plus surgical RV remodeling to PVR alone.

Research Question:

Is there a difference between two surgical strategies-PVR alone (bioprosthetic pulmonary valve insertion and, when present, resection of right ventricular outflow tract [RVOT] aneurysm) versus PVR and surgical RV remodeling (bioprosthetic pulmonary valve insertion and resection of akinetic scarred areas on the anterior RV wall to reduce RV volume)-on RV mechanics and on the incidence of adverse events in patients with repaired TOF and chronic pulmonary regurgitation?

ELIGIBILITY:
Inclusion Criteria:

* Undergoing PVR to repair TOF at Children's Hospital Boston
* Pulmonary regurgitation fraction greater than or equal to 25% (measured by CMR) and two or more of the following criteria:

  1. RV end-diastolic volume index greater than or equal to 150 ml/m2 (Z score greater than 5)
  2. RV end-systolic volume index greater than or equal to 70 ml/m2
  3. LV end-diastolic volume index less than or equal to 65 ml/m2
  4. RV ejection fraction less than 45%
  5. RVOT aneurysm
  6. Clinical criteria: exercise intolerance, symptoms and signs of heart failure, and use of cardiac medications

Exclusion Criteria:

* Presence of either severe RV outflow tract obstruction (defined as peak-to-peak systolic gradient of greater than or equal to 60 mm Hg by cardiac catheterization) or severe RV hypertension at systemic or higher level
* Additional sources of RV volume overload other than PR and tricuspid valve regurgitation
* Contraindications to CMR

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2004-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Changes in ventricular mechanics compared with the preoperative ventricular mechanics | Measured at 6 months

SECONDARY OUTCOMES:
Incidence of one or more postoperative adverse events | Measured at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tal Geva, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Department of Cardiology, Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Geva T, Gauvreau K, Powell AJ, Cecchin F, Rhodes J, Geva J, del Nido P. Randomized trial of pulmonary valve replacement with and without right ventricular remodeling surgery. Circulation. 2010 Sep 14;122(11 Suppl):S201-8. doi: 10.1161/CIRCULATIONAHA.110.951178. PMID 20837914